CLINICAL TRIAL: NCT04774744
Title: Evaluating the Effect of a Digital Coaching Program on Self-Efficacy and Patient Reported Outcomes of Individuals With Acute and Chronic Leukemia
Brief Title: Effect of Digital Health Coaching Program on Self-efficacy and Patient Reported Outcomes of Patients With Newly Diagnosed Acute Myeloid Leukemia or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0806; NCI-2020-07406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0806 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-10-14; First posted 2021-03-01 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Early Intervention, Educational; Educational Status; Methods; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (digital health coaching program) (Experimental): Patients receive the PACK Health digital health coaching program over 3 months consisting of communication initiated by either the PACK Health coach or the patient through either text, e-mail, or phone call, to provide education and support related to a specific topic such as fatigue, nutrition, or exercise.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration
- Group II (standard of care support services) (Active Comparator): Patients receive standard of care support services consisting of a telephone triage line that patients may call when experiencing physical or psychological concerns, or with any other questions related to their disease or treatment.
  Interventions: Other: Questionnaire Administration; Other: Supportive Care

INTERVENTIONS:
Other: Educational Intervention — Receive digital health coaching program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group I (digital health coaching program)
Other: Questionnaire Administration — Ancillary studies
Other: Supportive Care — Receive standard of care support services
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Group II (standard of care support services)

SUMMARY:
This trial studies the effect of a digital health coaching program on self-efficacy and patient reported outcomes of patients with acute myeloid leukemia or chronic lymphocytic leukemia that is newly diagnosed. A digital health coaching program may help leukemia patients report information about their health while receiving treatment, which may lead to improvement in overall health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of digital health coaching on self-efficacy among two cohorts of individuals with acute myeloid leukemia (AML) and chronic lymphocytic leukemia (CLL), respectively, as measured by the Cancer Behavior Inventory (CBI version [v.] 3).

SECONDARY OBJECTIVES:

I. To evaluate the relationship between self-efficacy and patient reported outcomes among individuals with and without digital health coaching, specifically:

Ia. The physiologic and psychosocial outcomes of individuals with AML and CLL as measured by the Functional Assessment of Cancer Therapy-Leukemia Questionnaire (FACT-Leu).

Ib. The symptom experience of individuals with AML and CLL as measured by the MD Anderson Symptom Inventory (MDASI).

Ic. The financial toxicity of individuals with AML and CLL as measured by the Comprehensive Score for Financial Toxicity (COST).

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive the PACK Health digital health coaching program over 3 months consisting of communication initiated by either the PACK Health coach or the patient through either text, e-mail, or phone call, to provide education and support related to a specific topic such as fatigue, nutrition, or exercise.

GROUP II: Patients receive standard of care support services consisting of a telephone triage line that patients may call when experiencing physical or psychological concerns, or with any other questions related to their disease or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, speak and consent in English
* Individuals newly diagnosed with either acute myelogenous (AML) or chronic lymphocytic leukemia (CLL), defined as within three months of diagnosis
* Internet access via smart phone, tablet, a computer, or another device with the capacity to receive calls, texts, or e-mails, as well as the electronic study assessments
* Individuals with a prior history of myelodysplastic syndrome (MDS) will be allowed to enroll

Exclusion Criteria:

* Individuals who are terminally ill, defined as individuals identified by their physician as likely having 6 months or less to live, or those individuals transitioned to comfort measures only (meaning only supportive care measures without curative focused treatment)
* Individuals who have undergone treatment for previous diagnoses of leukemia
* Individuals for whom there is documentation of inability to provide consent in the medical record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Cancer Behavior Inventory (CBI) score | Baseline to 3 months
  The Cancer Behavior Inventory (CBI) is 27-item instrument that measures self-efficacy in coping with cancer across 7 domains. These include: Seeking and Understanding Medical Information, Emotion Regulation, Coping with Treatment Related Side Effects, Accepting Cancer/ Maintaining a Positive Attitude, Seeking Social Support, and Using Spiritual Coping. The instrument utilizes a 7-point response scale ranging from 1 "Not at all confident" to 7 "Confident" (higher score equals greater efficacy for coping).
  * Minimum Score-27, max- 189
  * Will be calculated along with 95% confidence intervals.

SECONDARY OUTCOMES:
Physiologic and psychosocial outcomes | Up to 3 months
  Linear mixed models (LMMs) will be created to assess the correlation between self-efficacy, using the Cancer behavior inventory (CBI), and physiologic and psychosocial outcomes (as measured by the Functional Assessment of Cancer Therapy-Leukemia Questionnaire).
  The Functional Assessment of Cancer Therapy with Leukemia Questionnaire (FACT-Leu) is a 44-item measure of quality of life associated with leukemia treatment. It consists of 4 defined domains: physical, social, emotional, and functional, as well as 17 items related to additional disease and treatment related concerns. Responses are measured on a five-point scale ranging from 0 (not at all) to 4 (very much).
  • Minimum Score -0, Maximum Score - 176
Symptom experience | Up to 3 months
  Linear mixed models will be created to assess the correlation between self-efficacy (CBI) and symptom experience (as measured by the MD Anderson Symptom Inventory).
  The MD Anderson Symptom Inventory (MDASI) is a multiple-symptom measure of the severity of cancer-related symptoms and the functional interference caused by symptoms that is sensitive to disease and treatment changes. Patients rate the severity of 13 physical, affective, and cognitive symptoms on 0-10 numeric scales, ranging from "not present" to "as bad as you can imagine." The MDASI also assesses 6 items related to symptom interference with functioning, also a 0-10 numeric scale ranging from "did not interfere" to "interfere completely." The MDASI takes less than five minutes to complete.
  • Minimum Score - 0, Maximum Score - 190
Perceived financial toxicity | Up to 3 months
  LMMs will be created to assess the correlation between self-efficacy (CBI) and perceived financial toxicity (as measured by the Comprehensive Score for Financial Toxicity).
  Comprehensive Score for Financial Toxicity (COST) is an 11-item instrument used to measure the financial toxicity of cancer treatment, which has been demonstrated to be highly correlated with HRQoL. The instrument consists of 11 items, utilizing a five-point ordinal scale ranging from (0- Not at all) to (4- Very much).
  • Minimum Score - 12, Maximum Score - 28

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org